CLINICAL TRIAL: NCT03670810
Title: Randomized Controlled Trial of Lasmiditan Over Four Migraine Attacks
Brief Title: A Study of Lasmiditan (LY573144) Over Four Migraine Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17131; H8H-MC-LAIJ (Other: Eli Lilly and Company); 2018-001661-17 (EudraCT Number)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-06

CONDITIONS: Migraine
Keywords: acute treatment; migraine pain; multiple attacks; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- 100 milligram (mg) Lasmiditan (Experimental): Participants received one 100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100 mg Lasmiditan matching placebo tablet to maintain blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- 200 mg Lasmiditan (Experimental): Participants received two 100 mg Lasmiditan tablets with one 50 mg Lasmiditan matching placebo tablet to maintain blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- Control 1 Sequence (Placebo Comparator): Control 1:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- Control 2 Sequence (Placebo Comparator): Control 2:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attack 4.
  Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- 100 mg Lasmiditan Maximum Extended Enrollment (MEE) (Experimental): Participants received one 100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100 mg Lasmiditan matching placebo tablet to maintain blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- 200 mg Lasmiditan MEE (Experimental): Participants received two 100 mg Lasmiditan tablets with one 50 mg Lasmiditan matching placebo tablet to maintain blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- Control 1 Sequence MEE (Placebo Comparator): Control 1:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- Control 2 Sequence MEE (Placebo Comparator): Control 2:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 4.
  Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- Open Label Extension (Experimental): Participants initially received 100 mg Lasmiditan at the first OLE visit, with flexible dosing (50, 100, or 200 mg) thereafter to optimize efficacy and tolerability.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally.
  Other Names: LY573144
Drug: Placebo — Administered orally.
  Arms: 100 mg Lasmiditan Maximum Extended Enrollment (MEE); 100 milligram (mg) Lasmiditan; 200 mg Lasmiditan; 200 mg Lasmiditan MEE; Control 1 Sequence; Control 1 Sequence MEE; Control 2 Sequence; Control 2 Sequence MEE

SUMMARY:
The reason for this study is to see how effective and safe the study drug known as lasmiditan is in the acute treatment of 4 migraine attacks with or without aura.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura fulfilling the International Headache Society (IHS) diagnostic criteria 1.1 and 1.2.1
* History of disabling migraine for at least 1 year
* Migraine onset before the age of 50 years
* History of 3 to 8 migraine attacks per month (<15 headache days per month) during the past 3 months
* MIDAS score ≥11
* Able and willing to complete an eDiary to record the details of each migraine attack treated with study drug
* Women of child-bearing potential must be using or willing to use a highly effective form of contraception
* Agree not to post any personal medical data or information related to the study on any website or social media site until the entire trial has completed

Exclusion Criteria:

* Known hypersensitivity to lasmiditan, or to any excipient of lasmiditan oral tablets
* History or evidence of hemorrhagic stroke, epilepsy, or any other condition placing the participant at increased risk of seizures
* History of recurrent dizziness and/or vertigo including benign paroxysmal positional vertigo, Meniere's disease, vestibular migraine, and other vestibular disorders
* History of diabetes mellitus with complications (diabetic retinopathy, nephropathy, or neuropathy)
* History of orthostatic hypotension with syncope
* Significant renal or hepatic impairment in the opinion of the investigator or if they meet hepatic monitoring criteria
* Participants who, in the investigator's judgment, are actively suicidal and therefore deemed to be at significant risk for suicide
* History, within past 12 months, of chronic migraine or other forms of primary or secondary chronic headache disorder (eg, hemicranias continua, medication overuse headache where headache frequency is ≥15 headache days per month)
* Use of more than 3 doses per month of either opioids or barbiturates
* Initiation of or a change in concomitant medication to reduce the frequency of migraine episodes within 3 months prior to screening
* Pregnant or breast-feeding women
* History of drug or alcohol abuse/dependence within 1 year prior to screening
* Any medical condition or clinical laboratory test which in the judgment of the investigator makes the participant unsuitable for the study
* Currently enrolled in any other clinical study involving an investigational product
* Relatives of, or staff directly reporting to, the Investigator
* Participants who are employees of the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1633 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (141):
- United States (14):
  - Rehabilitation & Neurological Services LLC, Huntsville, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - UCSD Altman Clinical & Translational Research Institute (ACTRI), La Jolla, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Diamond Headache Clinic, Chicago, Illinois
  - Ochsner Medical Center - North Shore, Covington, Louisiana
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Nevada Headache Institute, Las Vegas, Nevada
  - Dent Neurological Institute, Amherst, New York
  - Island Neuro Associates,PC, Plainview, New York
  - Montefiore Headache Center, The Bronx, New York
  - Northwest Clinical Research Center, Bellevue, Washington
- Austria (4):
  - Universitätsklinik Innsbruck, Innsbruck, Tyrol
  - KH der Barmherzigen Schwestern Linz BetriebsGesmbH, Linz, Upper Austria
  - Christian-Doppler-Klinik, Salzburg
  - AKH, Vienna
- Belgium (6):
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Algemeen Ziekenhuis St Jan Brugge, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - CHC MontLégia, Liège
  - Valdor - ISOSL CCV - Clinique des céphalées du Valdor - Neurology, Liège
- China (29):
  - Beijing Tiantan Hospital Affiliated to Capital Medical Univ, Beijing, Beijing Municipality
  - Xuanwu Hospital-Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - First hospital affiliated to Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union (Xiehe) Hospital, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - People's hospital of Rizhao, Rizhao, Shandong
  - HuaShan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - No 1 Affiliate Hospital of Kunming Medical College, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Baotou Central Hospital, Baotou
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Tianjin Medical University General Hospital, Tianjin
- Czechia (6):
  - Clintrial, s.r.o., Prague, Hl. M. Praha
  - Neurologicka ambulance, Neurologie Brno s.r.o., Brno
  - Brain-Soultherapy s.r.o, Kladno
  - DADO MEDICAL, s.r.o., Prague
  - Neurologicka ordinace, Prague
  - Neurologicka ambulance Prerov, Přerov
- Denmark (3):
  - CCBR-Alborg-DK, Aalborg
  - Glostrup Hospital, Glostrup Municipality
  - Center for Clinical and Basic Research -CCBR, Vejle
- France (5):
  - APHM Hôpital de la Timone, Marseille
  - Centre Hospitalier Annecy Genevois - Site d'Annecy, Metz-Tessy
  - Hopital Lariboisière, Paris
  - CHU de Rouen Hopital Charles Nicolle, Rouen
  - CHU St Etienne Hopital Nord, Saint-Etienne
- Germany (13):
  - Synexus Clinical Research GmbH, Frankfurt am Main, Hesse
  - DRK-Kliniken Nordhessen, Kassel, Hesse
  - Gemeinschaftspraxis für Neurologie und Psychiatrie, Westerstede, Lower Saxony
  - Praxis Dr. Philipp Stude, Bochum, North Rhine-Westphalia
  - Synexus Clinical Research GmbH, Bochum, North Rhine-Westphalia
  - DataMed Klinische Studien GmbH, Cologne, North Rhine-Westphalia
  - Praxis für Neurologie und Psychiatrie, Essen, North Rhine-Westphalia
  - Synexus Clinical Research GmbH, Leipzig, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Neurologische Praxis Eppendorf, Hamburg
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
- Hungary (3):
  - Valeomed Kft., Esztergom, Komárom-Esztergom
  - SE Neurologiai Klinika, Budapest
  - Orszagos Idegtudomanyi Intezet, Budapest
- India (10):
  - Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Apollo Hospitals International Ltd., Ahmedabad, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - Mangala Hospitals & Mangala Kidney Foundation, Mangalore, Karnataka
  - Kokilaben Dhirubhai Ambani Hospital &Medical Research Inst., Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanth Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Gobind Ballabh Pant Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
- Italy (4):
  - Istituto Neurologico Neuromed, Pozzilli, Isernia
  - Ospedale Bellaria, Bologna
  - Istituto Neurologico Carlo Besta, Milan
  - Fondazione Istituto Neurologico Nationale C. Mondino, Pavia
- Mexico (8):
  - Clinical Research Institute S C, Tlalnepantla, Edo de Mex
  - Clinstile, S.A de C.V, Cuauhtémoc, Federal District
  - CRI Centro Regiomontano de Investigacion S.C., Monterrey, Nuevo León
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Medical Care and Research, S.A. de C.V., Mérida, Yucatán
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
  - Eci Estudios Clinicos Int., Puebla City
  - Centro de Atención e Investigación Cardiovascular del Potosí S.C., San Luis Potosí City
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Boerhaave Medisch Centrum, Amsterdam
  - Isala Klinieken, Zwolle
- Russia (4):
  - First Moscow State Medical University n.a. Sechenov, Moscow
  - University Headache Clinic, Moscow
  - Medis Priokskiy, Nizhny Novgorod
  - Saint Petersburg State Medical University n.a. Pavlov I.P., Saint Petersburg
- Spain (10):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - H.C.U. Lozano Blesa, Zaragoza
- Switzerland (5):
  - Kantonsspital Luzern, Lucerne, Canton of Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - KopfwehZentrum Hirslanden Zürich, Zollikon, Canton of Zurich
  - Rehaclinic Bad Zurzach, Bad Zurzach
  - Inselspital Bern, Bern
- United Kingdom (14):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Hull Royal Infirmary, Hull, East Yorkshire
  - Kings College Hospital, London, Greater London
  - Re-Cognition Health Ltd, London, Greater London
  - Synexus Manchester Clinical Research Centre, Manchester, Greater Manchester
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus Merseyside Clinical Research Centre, Liverpool, Merseyside
  - Synexus Hexham General Hospital, Hexham, Northumberland
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Synexus Wales Clinical Research Centre, Cardiff, South Glamorgan
  - Synexus Scotland Clinical Research Centre, Glasgow, Strathclyde
  - Re-Cognition Health Ltd, Guildford, Surrey
  - Re-Cognition Health Ltd, Birmingham, West Midlands
  - Synexus Midlands Clinical Research Center, Birmingham, Wstmid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Komori M, Ozeki A, Tanji Y, Kamiki E, Krege JH, Li LQ, Suzuki S, Shibata M, Takeshima T. Long-term treatment with lasmiditan in patients with migraine: post hoc analysis of treatment patterns and outcomes from the open-label extension of the CENTURION randomized trial. J Headache Pain. 2024 Mar 25;25(1):43. doi: 10.1186/s10194-024-01745-y. PMID 38528476
- [Derived] Blumenfeld A, Tepper SJ, Khanna R, Doty E, Vincent M, Miller SI. Serotonin syndrome in the acute treatment landscape of migraine: the lasmiditan experience. Front Neurol. 2023 Oct 27;14:1291102. doi: 10.3389/fneur.2023.1291102. eCollection 2023. PMID 37965170
- [Derived] Ashina M, Roos C, Li LQ, Komori M, Ayer D, Ruff D, Krege JH. Long-term treatment with lasmiditan in patients with migraine: Results from the open-label extension of the CENTURION randomized trial. Cephalalgia. 2023 Apr;43(4):3331024231161745. doi: 10.1177/03331024231161745. PMID 36950929
- [Derived] Zhou J, Luo G, Xu Y, Yang X, Pan X, Dong Z, Zhong S, Liu H, Ji F, Yu S. Safety Findings in Lasmiditan as a Novel Acute Treatment of Migraine in Chinese Patients: A Post Hoc Analysis of the Randomized Controlled Phase 3 CENTURION Trial. Adv Ther. 2022 Nov;39(11):5229-5243. doi: 10.1007/s12325-022-02291-2. Epub 2022 Sep 17. PMID 36114949
- [Derived] MacGregor EA, Komori M, Krege JH, Baygani S, Vincent M, Pavlovic J, Igarashi H. Efficacy of lasmiditan for the acute treatment of perimenstrual migraine. Cephalalgia. 2022 Dec;42(14):1467-1475. doi: 10.1177/03331024221118929. Epub 2022 Aug 18. PMID 35979677
- [Derived] Doty EG, Hauck PM, Krege JH, Komori M, Hake AM, Dong Y, Lipton RB. The Association Between the Occurrence of Common Treatment-Emergent Adverse Events and Efficacy Outcomes After Lasmiditan Treatment of a Single Migraine Attack: Secondary Analyses from Four Pooled Randomized Clinical Trials. CNS Drugs. 2022 Jul;36(7):771-783. doi: 10.1007/s40263-022-00928-y. Epub 2022 Jul 2. PMID 35779194
- [Derived] Yu T, He L, Yang X, Zhou J, Luo G, Wang H, Zhao H, Hu Q, Ji F, Yu S. Efficacy and Safety of Lasmiditan as a Novel Acute Treatment in Chinese Patients with Migraine: A Subpopulation Analysis of the Randomized Controlled Phase 3 CENTURION Trial. Neurol Ther. 2022 Sep;11(3):1269-1283. doi: 10.1007/s40120-022-00369-1. Epub 2022 Jun 17. PMID 35713760
- [Derived] Krege JH, Lipton RB, Baygani SK, Komori M, Ryan SM, Vincent M. Lasmiditan for Patients with Migraine and Contraindications to Triptans: A Post Hoc Analysis. Pain Ther. 2022 Jun;11(2):701-712. doi: 10.1007/s40122-022-00388-8. Epub 2022 Apr 26. PMID 35471625
- [Derived] Tassorelli C, Bragg S, Krege JH, Doty EG, Ardayfio PA, Ruff D, Dowsett SA, Schwedt T. Safety findings from CENTURION, a phase 3 consistency study of lasmiditan for the acute treatment of migraine. J Headache Pain. 2021 Nov 6;22(1):132. doi: 10.1186/s10194-021-01343-2. PMID 34742230
- [Derived] Reuter U, Krege JH, Lombard L, Gomez Valderas E, Krikke-Workel J, Dell-Agnello G, Dowsett SA, Buse DC. Lasmiditan efficacy in the acute treatment of migraine was independent of prior response to triptans: Findings from the CENTURION study. Cephalalgia. 2022 Jan;42(1):20-30. doi: 10.1177/03331024211048507. Epub 2021 Oct 13. PMID 34644189
- [Derived] Ashina M, Reuter U, Smith T, Krikke-Workel J, Klise SR, Bragg S, Doty EG, Dowsett SA, Lin Q, Krege JH. Randomized, controlled trial of lasmiditan over four migraine attacks: Findings from the CENTURION study. Cephalalgia. 2021 Mar;41(3):294-304. doi: 10.1177/0333102421989232. Epub 2021 Feb 4. PMID 33541117
- See also: A Study of Lasmiditan (LY573144) Over Four Migraine Attacks — https://trials.lillytrialguide.com/en-US/trial/45cVxLjssEICmyC0uECUa4

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were considered study completers after treating 4 migraine attacks or after completing 4 months of study duration regardless of number of treated attacks in the main study. Participants may continue in Open-Label Extension (OLE) if they met OLE eligibility criteria.
Pre-assignment Details: An ITT evaluable attack is defined as a treated attack of least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose.
Groups:
- 100 Milligram (mg) Lasmiditan: Participants received one100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100-mg Lasmiditan matching placebo tablet to maintain blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
- 100 mg Lasmiditan Maximum Extended Enrollment (MEE): Participants received one100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100 mg Lasmiditan matching placebo tablet to maintain blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
- Control 2 Sequence MEE: Control 2:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attack 4.
  Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
- Open-Label Extension: Participants initially received 100 mg Lasmiditan at the first OLE visit, with flexible dosing (50, 100, or 200 mg) thereafter to optimize efficacy and tolerability.
Period: Main Study
Arm/Group | 100 Milligram (mg) Lasmiditan | 200 mg Lasmiditan | Control 1 Sequence | Control 2 Sequence | 100 mg Lasmiditan Maximum Extended Enrollment (MEE) | 200 mg Lasmiditan MEE | Control 1 Sequence MEE | Control 2 Sequence MEE | Open-Label Extension
Started | 485 | 486 | 249 | 251 | 55 | 53 | 28 | 26 | 0
Treated at Least One Migraine Attack | 485 | 486 | 249 | 251 | 55 | 53 | 28 | 26 | 0
Completed | 403 | 394 | 219 | 223 | 45 | 46 | 26 | 23 | 0
Not Completed | 82 | 92 | 30 | 28 | 10 | 7 | 2 | 3 | 0
Not completed — Adverse Event | 37 | 38 | 3 | 4 | 4 | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 9 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 7 | 4 | 6 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Pregnancy | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 2 | 12 | 8 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 21 | 8 | 9 | 5 | 2 | 1 | 1 | 0
Not completed — Participant did not want to take the three other treatments | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Migraines more frequent-GP advised to re-start Topiramate | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Travel and Coronavirus issues | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open Label Extension
Arm/Group | 100 Milligram (mg) Lasmiditan | 200 mg Lasmiditan | Control 1 Sequence | Control 2 Sequence | 100 mg Lasmiditan Maximum Extended Enrollment (MEE) | 200 mg Lasmiditan MEE | Control 1 Sequence MEE | Control 2 Sequence MEE | Open-Label Extension
Started | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 0 (Reported are only those participants who were enrolled in the OLE.) | 477
Treated at Least One Migraine Attack | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 476 (One participant signed consent but decided against participating in the OLE period and was not dosed.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 324
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 153
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — COVID-19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39
Not completed — Participant refused to comply with face mask use | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Taking medication too restrictive for lifestyle | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46
Not completed — Participant didn't have disposition for OLE period | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
Not completed — Participant wanted to become pregnant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23

BASELINE CHARACTERISTICS:
Population: All randomized participants who were treated with at least 1 dose of study drug, regardless of whether or not they undergo any study assessments.
Groups:
- 100 mg Lasmiditan: Participants received one 100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100 mg Lasmiditan matching placebo tablet to maintain blind.
- 200 mg Lasmiditan: Participants received two 100 mg Lasmiditan tablets with one 50 mg Lasmiditan matching placebo tablet to maintain blind.
- Control: Control 1: Participants received one 50 mg Lasmiditan matching placebo tablet and two100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4.
  Participants received one50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Control 2: Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to treat migraine attacks 1, 2 and 3.
  Participants received one 50 mg Lasmiditan tablet and two 100 mg Lasmiditan matching placebo tablets to treat migraine attack 4.
- 100 mg Lasmiditan MEE: Participants received one 100 mg Lasmiditan tables with one 50 mg lasmiditan matching placebo tablet and one 100 mg Lasmiditan matching placebo tablet to maintain the blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
- 200 mg Lasmiditan MEE: Participants received two 100 mg Lasmiditan tables with one 50 mg lasmiditan matching placebo tablet to maintain the blind. Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
- Control MEE: Control 1:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Control 2:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attack 4.
  Tablets were administered orally within 4 hours of onset of a single migraine attack, up to 4 migraine attacks.
- Total: Total of all reporting groups
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Control | 100 mg Lasmiditan MEE | 200 mg Lasmiditan MEE | Control MEE | Total
Number analyzed (Participants) | 485 | 486 | 500 | 55 | 53 | 54 | 1633
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.90 (12.02) | 41.70 (11.95) | 40.60 (12.11) | 37.20 (9.83) | 37.20 (9.46) | 38.60 (8.70) | 41.30 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 403 | 418 | 416 | 43 | 36 | 40 | 1356
  Male | 82 | 68 | 84 | 12 | 17 | 14 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 44 | 47 | 0 | 0 | 0 | 135
  Not Hispanic or Latino | 393 | 390 | 401 | 19 | 14 | 15 | 1232
  Unknown or Not Reported | 48 | 52 | 52 | 36 | 39 | 39 | 266
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 25 | 28 | 27 | 0 | 0 | 0 | 80
  Asian | 71 | 72 | 78 | 53 | 49 | 51 | 374
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 12 | 8 | 7 | 0 | 0 | 0 | 27
  White | 370 | 368 | 379 | 2 | 4 | 3 | 1126
  More than one race | 0 | 2 | 1 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 7 | 7 | 8 | 0 | 0 | 0 | 22
Region of Enrollment [Number; unit: participants]
  Austria | 5 | 3 | 3 | 0 | 0 | 0 | 11
  Belgium | 9 | 10 | 9 | 0 | 0 | 0 | 28
  China | 45 | 44 | 47 | 50 | 48 | 47 | 281
  Czechia | 33 | 32 | 31 | 0 | 0 | 0 | 96
  Denmark | 9 | 10 | 11 | 0 | 0 | 0 | 30
  France | 7 | 7 | 8 | 0 | 0 | 0 | 22
  Germany | 92 | 89 | 94 | 0 | 0 | 0 | 275
  Hungary | 6 | 6 | 5 | 0 | 0 | 0 | 17
  India | 12 | 14 | 13 | 3 | 1 | 4 | 47
  Italy | 7 | 7 | 8 | 0 | 0 | 0 | 22
  Mexico | 29 | 32 | 34 | 0 | 0 | 0 | 95
  Netherlands | 3 | 4 | 3 | 0 | 0 | 0 | 10
  Russia | 13 | 12 | 13 | 2 | 4 | 3 | 47
  Spain | 18 | 21 | 22 | 0 | 0 | 0 | 61
  Switzerland | 5 | 7 | 7 | 0 | 0 | 0 | 19
  United Kingdom | 164 | 162 | 164 | 0 | 0 | 0 | 490
  United States | 28 | 26 | 28 | 0 | 0 | 0 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Are Pain Free 2 Hours Postdose During the First Attack
Description: Pain-free is defined as mild, moderate, or severe headache pain becoming none at 2 hours postdose during the first attack.
Time Frame: 2 Hours Postdose
Population: All randomized participants who used at least 1 dose of study drug for an Intent-to-Treat (ITT) evaluable attack, defined as a treated attack of at least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Groups:
- 100 mg Lasmiditan: Participants received one100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100-mg Lasmiditan matching placebo tablet to maintain blind.
- Placebo: Control 1:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Control 2:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attack 4.
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 25.8 | 29.3 | 8.4
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.83, 95% CI 2-sided [2.56 to 5.73]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.56, 95% CI 2-sided [3.07 to 6.77]

2. Primary Outcome: Percentage of Participants That Are Pain Free at 2 Hours Postdose in at Least 2 Out of 3 Attacks
Description: To evaluate the 2 out of 3 primary consistency endpoint, the results of ITT evaluable attacks in the lasmiditan 100-mg and 200-mg groups will be assessed, and the ITT-evaluable attacks treated with placebo in the control group will be used for comparison. For participants with more than 3 ITT evaluable attacks, only the first 3 will be considered. Pain-free was defined as mild, moderate, or severe headache pain becoming none at the indicated assessment time.
Time Frame: 2 Hours Postdose
Population: All randomized participants who experienced at least 2 successes or 2 failures during their first 2 or 3 ITT evaluable attacks. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 340 | 336 | 373
percentage of participants | 14.4 | 24.4 | 4.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 3.77, 95% CI 2-sided [2.10 to 6.76]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 7.24, 95% CI 2-sided [4.13 to 12.67]

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post Dose During the First Attack
Description: Headache pain-relief is defined as a reduction in pain severity from moderate or severe at baseline to mild or none, or a reduction in pain severity from mild at baseline to none, at the indicated assessment time.
Time Frame: 2 Hours Postdose
Population: All randomized participants who use at least 1 dose of study drug for an ITT evaluable attack, defined as a treated attack of at least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 65.4 | 65.2 | 41.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.71, 95% CI 2-sided [2.05 to 3.57]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [2.04 to 3.53]

4. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Postdose in at Least 2 Out of 3 Attacks
Description: Headache pain relief is defined as a reduction in pain severity from moderate to severe at baseline to mild or none at 2 hours postdose in at least 2 out of 3 attacks. To evaluate at least 2 out of 3 consistency endpoints, the results of ITT-evaluable attacks in the lasmiditan 100-mg and 200-mg groups will be assessed, and the ITT-evaluable attacks treated with placebo in the control group will be used for comparison. For participants with more than 3 ITT-evaluable attacks, only the first 3 with the same treatment will be considered.
Time Frame: 2 Hours Postdose
Population: All randomized participants who experienced a sufficient number of successes or failures, (2 successes or 2 failures ) during their first 2 or 3 ITT-evaluable attacks. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Groups:
- 100 mg Lasmiditan: Participants received one 100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100-mg Lasmiditan matching placebo tablet to maintain blind.
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 332 | 333 | 320
percentage of participants | 62.3 | 66.7 | 36.9
Statistical Analysis 1: Comparison: 100 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.91, 95% CI 2-sided [2.11 to 4.01]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.50, 95% CI 2-sided [2.53 to 4.85]

5. Secondary Outcome: Percentage of Participants With 24-Hour Sustained Pain Freedom During the First Attack
Description: Sustained pain freedom defined as pain free at 2 and 24 hours with no rescue medication.
Time Frame: 24 Hours
Population: All randomized participants who received at least 1 dose of study drug for an ITT evaluable attack, defined as a treated attack of at least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 13.6 | 17.3 | 4.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.52, 95% CI 2-sided [2.05 to 6.02]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.67, 95% CI 2-sided [2.77 to 7.88]

6. Secondary Outcome: Percentage of Participants With 48-Hour Sustained Pain Freedom During First Attack
Description: Sustained pain freedom defined as pain free at 2 and 48 hours with no rescue medication.
Time Frame: 48 Hours Postdose
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 9.3 | 15.4 | 4.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.30 to 4.04]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.09, 95% CI 2-sided [2.41 to 6.94]

7. Secondary Outcome: Percentage of Participants That Are Pain Free 2 Hours Postdose During the First Attack in Triptan Insufficient Responders.
Description: Pain-free is defined as mild, moderate, or severe headache pain becoming none at 2 hours postdose during the first attack. A triptan insufficient responder is defined as having one of the following: 1) Scoring ≤5 on 4 questions from the Migraine Treatment Optimization Questionnaire (mTOQ-6) that defines participants with poor or very poor response to their current regimen; 2) Indicated they obtained pain freedom at 2 hours in 0 out of 3, or 1 out of 3 attacks when treated with the most recent triptan, or 3) are not currently taking triptan and discontinued their most recent triptan due to lack of efficacy, tolerability issue, or contradictions to a past triptan.
Time Frame: 2 Hours Postdose
Population: All randomized participants who were triptan insufficient responders and used at least 1 dose of study drug for an ITT evaluable attack, defined as a treated attack of at least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 183 | 203 | 193
percentage of participants | 24.0 | 25.6 | 8.8
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.80 to 6.02]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.56, 95% CI 2-sided [1.97 to 6.42]

8. Secondary Outcome: Percentage of Participants With no Disability as Measured by the Disability Item, at 2 Hours Postdose During the First Attack
Description: Percentage of participants with no disability as measured by the disability item, at 2 hours postdose during the first attack. Disability was measured by determining the level of interference with normal activities with 4 response options including not at all; mild interference, marked interference; and need complete bed rest.
Time Frame: 2 Hours Postdose
Population: All randomized participants who used at least 1 dose of study drug for an ITT evaluable attack, defined as a treated attack of at least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 18.6 | 19.8 | 9.5
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.22, 95% CI 2-sided [1.48 to 3.33]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.46, 95% CI 2-sided [1.65 to 3.67]

9. Secondary Outcome: Percentage of Participants That Are Pain Free at 2 Hours Postdose in at Least 2 Out of 3 Attacks in Triptan Insufficient Responders
Description: Headache pain-free is defined as a reduction in pain severity from mild, moderate, or severe at baseline to none at the indicated assessment time. A subject is not counted as being pain-free at a specific time point if she or he used rescue or recurrence medication at or before the specific time point.
Time Frame: 2 Hours Postdose
Population: All randomized participants who were triptan insufficient responders and experienced a sufficient number of successes or failures, (2 successes or 2 failures ) during their first 2 or 3 ITT-evaluable attacks. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 17 | 31 | 7
percentage of participants | 11.0 | 20.1 | 4.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.10 to 6.78]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.64, 95% CI 2-sided [2.40 to 13.25]

10. Secondary Outcome: Percentage of Participants Free of Most Bothersome Symptom (MBS) Associated With Migraine at 2 Hours Postdose During the First Attack
Description: MBS freedom is defined as the absence of the associated symptom of migraine (nausea, phonophobia, or photophobia) at the indicated assessment time that was identified at baseline as the most bothersome symptom.
Time Frame: 2 Hours Postdose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 376 | 395 | 396
percentage of participants | 40.4 | 39.0 | 28.0
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.29 to 2.35]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.21 to 2.20]

11. Secondary Outcome: Percentage of Participants Requiring Rescue Medication for Migraine Within 24 Hours of Treatment During the First Attack
Description: Percentage of participants requiring rescue medication for migraine within 2 to 24 hours of treatment during the first attack
Time Frame: 24 Hours
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 311 | 307 | 406
percentage of participants | 19.6 | 19.2 | 29.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.33 to 0.65]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.30 to 0.60]

12. Secondary Outcome: Percentage of Participants That Are Free of Symptoms Associated With Migraine at 2 Hours Postdose During the First Attack
Description: Percentage of participants that are free of symptoms associated with migraine (photophobia, phonophobia, nausea, and vomiting) at 2 hours postdose during the first attack.
Time Frame: 2 Hours Postdose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 17.9 | 21.0 | 7.2
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.79 to 4.28]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.37, 95% CI 2-sided [2.20 to 5.15]

13. Secondary Outcome: Percentage of Participants With Migraine Recurrence at 24 Hours During the First Attack
Description: Percentage of participants with migraine recurrence at 24 hours during the first attack defined as return of any headache in participants who were pain free at 2 hours.
Time Frame: 24 Hours
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 108 | 127 | 37
percentage of participants | 30.6 | 22.0 | 37.8

14. Secondary Outcome: Percentage of Participants With Pain Freedom, Pain Relief, Freedom From MBS, and No Disability Postdose During First Attack
Description: Percentage of participants with pain freedom, pain relief, freedom from MBS, and no disability postdose during first attack.
Time Frame: 30 Minutes (Min) and 1 Hour (Hr) Postdose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants
  Pain Freedom (30 Min) | 1.4 | 1.6 | 0.2
  Pain Freedom (1Hr) | 6.0 | 12.7 | 2.0
  Pain Relief (30 Min) | 18.6 | 22.4 | 14.0
  Pain Relief (1 Hr) | 48.7 | 47.2 | 29.3
  Freedom from MBS (30 Min) | 12.5 | 14.4 | 11.4
  Freedom from MBS (1 Hr) | 23.7 | 28.9 | 22.0
  No Disability Postdose During First Attack (30 Min) | 3.1 | 2.3 | 2.3
  No Disability Postdose During First Attack (1 Hr) | 6.0 | 9.9 | 5.0
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Pain Freedom 30 Min. Postdose; Test type: Superiority; p = 0.086, Regression, Logistic; Odds Ratio (OR) = 6.40, 95% CI 2-sided [0.77 to 53.37]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Pain Freedom 30 Min. Postdose; Test type: Superiority; p = 0.065, Regression, Logistic; Odds Ratio (OR) = 7.24, 95% CI 2-sided [0.89 to 59.08]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; Pain Free 1 Hour Postdose; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.42 to 6.68]
Statistical Analysis 4: Comparison: 200 mg Lasmiditan vs Placebo; Pain Free 1 Hour Postdose; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.04, 95% CI 2-sided [3.43 to 14.44]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; Pain Relief 30 Min Postdose 100 mg; Test type: Superiority; p = 0.065, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.98 to 2.03]
Statistical Analysis 6: Comparison: 200 mg Lasmiditan vs Placebo; Pain Relief 30 Min. Postdose 200 mg; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.25 to 2.52]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; Pain Relief 1 Hour Postdose 100 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.74 to 3.06]
Statistical Analysis 8: Comparison: 200 mg Lasmiditan vs Placebo; Pain Relief 1 Hour Postdose 200 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.64 to 2.88]
Statistical Analysis 9: Comparison: 100 mg Lasmiditan vs Placebo; Freedom from MBS 30 Min 100 mg; Test type: Superiority; p = 0.651, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.71 to 1.71]
Statistical Analysis 10: Comparison: 200 mg Lasmiditan vs Placebo; Freedom from MBS 30 Min. 200 mg; Test type: Superiority; p = 0.220, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.85 to 1.98]
Statistical Analysis 11: Comparison: 100 mg Lasmiditan vs Placebo; Freedom from MBS 1 Hour 100 mg; Test type: Superiority; p = 0.593, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.78 to 1.54]
Statistical Analysis 12: Comparison: 200 mg Lasmiditan vs Placebo; Freedom from MBS 1 Hour 200 mg; Test type: Superiority; p = 0.030, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.04 to 1.98]

15. Secondary Outcome: Change From Baseline in Total Score as Measured by the Migraine Disability Assessment Test (MIDAS) Scale
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of 5 items that reflect the number of days reported as missed, or with reduced productivity at work or home and social events. Each question is answered as the number of days during the past 3 months of assessment, ranging from 0 to 90, with the total score being the summation of the 5 numeric responses. A higher value is indicative of more disability.
Time Frame: Baseline, Week 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Control 1:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Control 2:
  Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3.
  Participants received one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attack 4.
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Control
Number analyzed (Participants) | 447 | 437 | 451
score on a scale | -10.7 (24.36) | -12.0 (21.38) | -13.1 (21.40)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Control; Test type: Superiority; p = 0.092, ANCOVA
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Control; Test type: Superiority; p = 0.211, ANCOVA

16. Secondary Outcome: Percentage of Participants Very Much or Much Better as Measured by Patient Global Impression of Change (PGI-C), at 2 Hours Postdose During the First Attack
Description: The PGI-C is a one-item questionnaire that asks participants to provide their impression of change since taking the medicine. The PGI-C is measured using a 7-point Likert scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse. Reported are participants whose combined impression of change since taking the medicine was very much better and much better at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants | 29.8 | 30.0 | 13.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.85, 95% CI 2-sided [2.01 to 4.05]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.00, 95% CI 2-sided [2.12 to 4.26]

17. Secondary Outcome: Migraine Quality of Life Questionnaire (MQoLQ) Score at 24 Hours Post First Dose of Study During First Attack
Description: The 24-hour Migraine Quality of Life Questionnaire (24-hr MQoLQ) has been specifically developed to measure the HRQoL of participants with migraine within a 24-hour period after having taken migraine medication A domain score is calculated by summing the responses to the 3 questions and the domain score ranges from 3 to 21, with lower scores indicating less impairment. The questionnaire will be administered 24 hours after dosing with study drug during each migraine. The analysis of variance (ANOVA) model was used with region and treatment adjusted for the overall treatment effect.
Time Frame: 24 Hours Post First Dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 289 | 303 | 293
score on a scale
  Social Functioning | 12.4 (4.8) | 12.1 (4.7) | 11.7 (4.7)
  Migraine Symptoms | 12.4 (4.1) | 12.5 (4.2) | 11.4 (4.4)
  Feeling/Concern | 11.2 (4.3) | 11.2 (4.5) | 10.3 (4.2)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Social Functioning; Test type: Superiority; p = 0.056, ANOVA
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Social Functioning; Test type: Superiority; p = 0.267, ANOVA
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; Migraine Symptoms 100 mg; Test type: Superiority; p = 0.003, ANOVA
Statistical Analysis 4: Comparison: 200 mg Lasmiditan vs Placebo; Migraine Symptoms 200 mg; Test type: Superiority; p = 0.002, ANOVA
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; Feeling/Concerns 100 mg; Test type: Superiority; p = 0.014, ANOVA
Statistical Analysis 6: Comparison: 200 mg Lasmiditan vs Placebo; Feelings/Concerns 200 mg; Test type: Superiority; p = 0.018, ANOVA

18. Secondary Outcome: Percentage of Participants Satisfied With Their Treatment Measured by a 4-Item Questionnaire
Description: Treatment satisfaction was evaluated at the End of Study (EoS) visit by determining the participant's level of satisfaction (ranging from extremely dissatisfied to extremely satisfied); their willingness to take this treatment again (ranging from strongly disagree to strongly agree) and if they would they recommend this treatment to another participants (ranging from strongly disagree to strongly agree).
Time Frame: Week 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Control
Number analyzed (Participants) | 452 | 444 | 460
percentage of participants
  Recommend Treatment - Agree/Strongly Agree: number analyzed (Participants) | 451 | 444 | 460
  Recommend Treatment - Agree/Strongly Agree | 57.2 | 58.1 | 52.0
  Willing to Take Treatment - Agree/Strongly Agree | 61.5 | 58.9 | 64.3
  Extremely/Very Satisfied/Satisfied with Medication | 48.9 | 51.6 | 43.5
  Prefer This Treatment: number analyzed (Participants) | 141 | 145 | 134
  Prefer This Treatment | 31.2 | 32.7 | 29.1
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Control; Recommend Treatment - Agree Strongly Agree; Test type: Superiority; p = 0.101, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.96 to 1.62]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Control; Recommend Treatment Agree/Strongly Agree; Test type: Superiority; p = 0.063, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.67]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Control; Willing to Take This Treatment Again - Agree/Strongly Agree; Test type: Superiority; p = 0.376, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.68 to 1.16]
Statistical Analysis 4: Comparison: 200 mg Lasmiditan vs Control; Willing to Take This Treatment Again - Agree/Strongly Agree; Test type: Superiority; p = 0.082, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.60 to 1.03]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Control; Extremely/Very Satisfied; Test type: Superiority; p = 0.096, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.96 to 1.62]
Statistical Analysis 6: Comparison: 200 mg Lasmiditan vs Control; Extremely/Very Satisfied; Test type: Superiority; p = 0.016, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.06 to 1.80]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Control; Prefer This Treatment; Test type: Superiority; p = 0.445, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.84 to 1.49]
Statistical Analysis 8: Comparison: 200 mg Lasmiditan vs Control; Test type: Superiority; p = 0.243, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.89 to 1.58]

19. Secondary Outcome: Change From Baseline in Utility at 24 Hours Postdose as Measured by the EuroQol 5-Dimension 5-Level Scale (EQ-5D-5L) at 24 Hours Postdose During First Attack
Description: The EQ-5D-5L questionnaire is a participant-rated scale that assesses health status, it consists of 2 parts. The first part assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that have 5 possible levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems).The EQ-5D can be used to generate a health state index score, which is used to compute quality-adjusted life years for utilization in health economic analyses. The health state index score is calculated based on the responses to the 5 dimensions, providing a single value on a scale from less than 0 (where 0 is a health state equivalent to death) to 1 (perfect health), with higher scores indicating better health utility. ANCOVA was used to assess the effect of Lasmiditan over placebo or control. The model includes fixed categorical effect of treatment and geographic region and baseline as covariate.
Time Frame: Baseline, 24 Hours Postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
score on a scale | 0.2499 (0.25788) | 0.2270 (0.29854) | 0.2122 (0.25729)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs 200 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.142, ANCOVA

20. Secondary Outcome: Percentage of Participants That Are Pain Free at 2 Hours Postdose in at Least 3 Out of 4 Attacks
Description: Headache pain-free is defined as a reduction in pain severity from mild, moderate, or severe to none at the indicated assessment time (2 hours postdose). To evaluate 3 out of 4 consistency endpoints; all ITT-evaluable attacks will be used. For the control group, the results of all ITT-evaluable attacks treated with lasmiditan 50 mg or placebo will be included. The control group is used for comparison. The population for 3 out of 4 consistency endpoints with sufficient number of successes or failures is defined as all participants who experienced at least 3 successes or 2 failures during ITT-evaluable attacks.
Time Frame: 2 Hours Postdose
Population: All randomized participants who experienced a sufficient number of successes or failures, (3 out of 4 attacks) during ITT evaluable attacks for any of the consistency analyses. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Control
Number analyzed (Participants) | 325 | 306 | 387
percentage of participants | 7.4 | 10.8 | 2.6
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Control; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 3.01, 95% CI 2-sided [1.42 to 6.40]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Control; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.58, 95% CI 2-sided [2.22 to 9.47]

21. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Postdose in at Least 3 Out of 4 Attacks
Description: Headache pain-relief is defined as a reduction in pain severity from moderate or severe at baseline to mild or none, or a reduction in pain severity from mild at baseline to none, at the indicated assessment time (2 hours postdose). To evaluate 3 out of 4 consistency endpoints; all ITT-evaluable attacks will be used. For the control group, the results of all ITT-evaluable attacks treated with lasmiditan 50 mg or placebo will be included. The control group is used for comparison. The population for 3 out of 4 consistency endpoints with sufficient number of successes or failures is defined as all participants who experienced at least 3 successes or 2 failures during ITT-evaluable attacks.
Time Frame: 2 Hours Postdose
Population: All randomized participants who experienced a sufficient number of successes or failures, (3 successes or 2 failures ) during ITT-evaluable attacks for any of the consistency analyses. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Control
Number analyzed (Participants) | 260 | 257 | 317
percentage of participants | 40.8 | 49.8 | 21.8
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Control; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.74 to 3.62]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Control; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.61, 95% CI 2-sided [2.50 to 5.20]

22. Secondary Outcome: Percentage of Participants With Associated Migraines Symptoms of Nausea, Vomiting, Photophobia, and Phonophobia Present at 2 Hours Postdose for First Attack
Description: Presence of associated migraine symptoms at 2 hours postdose at first migraine attack, including each of the following: phonophobia, photophobia, nausea, and vomiting.
Time Frame: 2 Hours Postdose
Population: All randomized participants who used at least 1 dose of study drug for an Intent-to-Treat (ITT) evaluable attack, defined as a treated attack of at least mild pain severity with any postdose pain severity assessments at or before 2 hours postdose. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 419 | 434 | 443
percentage of participants
  Nausea | 29.1 | 29.0 | 29.1
  Phonophobia | 26.7 | 23.5 | 40.6
  Photophobia | 38.2 | 39.9 | 55.3
  Vomiting | 1.2 | 3.0 | 2.7
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Nausea; Test type: Superiority; p = 0.953, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.75 to 1.36]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Nausea; Test type: Superiority; p = 0.768, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.78 to 1.41]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; Phonophobia; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.39 to 0.71]
Statistical Analysis 4: Comparison: 200 mg Lasmiditan vs Placebo; Phonophobia; Test type: Superiority; p < 0.001, Regression, Linear; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.34 to 0.62]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; Photophobia; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.36 to 0.63]
Statistical Analysis 6: Comparison: 200 mg Lasmiditan vs Placebo; Photophobia; Test type: Superiority; p < 0.001, Regression, Logistic; Median Difference (Net) = 0.53, 95% CI 2-sided [0.40 to 0.71]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; Vomiting; Test type: Superiority; p = 0.129, Regression, Logistic; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.17 to 1.25]
Statistical Analysis 8: Comparison: 200 mg Lasmiditan vs Placebo; Vomiting; Test type: Superiority; p = 0.769, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.52 to 2.43]

ADVERSE EVENTS:
Time Frame: Up to 16 months
Description: All randomized participants who take at least 1 dose of study drug, regardless of whether or not they undergo any study assessments. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- 100 Milligram (mg) Lasmiditan; 100 mg Lasmiditan - MEE: Participants received one 100 mg Lasmiditan tablet with one 50 mg Lasmiditan matching placebo tablet and one 100-mg Lasmiditan matching placebo tablet to maintain blind.
- Main - Control; MEE - Control: Control 1 Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 4, and one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind, for migraine attack 3.
  Control 2 Participants received one 50 mg Lasmiditan matching placebo tablet and two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attacks 1, 2, and 3, and one 50 mg Lasmiditan tablet with two 100 mg Lasmiditan matching placebo tablets to maintain blind for migraine attack 4.
- 200 mg Lasmiditan - MEE: Participants received two 100 mg Lasmiditan tablets with one 50 mg Lasmiditan matching placebo tablet to maintain blind.
Arm/Group | 100 Milligram (mg) Lasmiditan | 200 mg Lasmiditan | Main - Control | 100 mg Lasmiditan - MEE | 200 mg Lasmiditan - MEE | MEE - Control | Open Label Extension
All-Cause Mortality (participants affected / at risk) | 0/485 | 0/486 | 0/500 | 0/55 | 0/53 | 0/54 | 1/477
Serious Adverse Events (participants affected / at risk) | 7/485 | 8/486 | 7/500 | 1/55 | 0/53 | 0/54 | 19/477
Other Adverse Events (participants affected / at risk) | 331/485 | 355/486 | 184/500 | 31/55 | 40/53 | 16/54 | 326/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 100 Milligram (mg) Lasmiditan (N=485) | 200 mg Lasmiditan (N=486) | Main - Control (N=500) | 100 mg Lasmiditan - MEE (N=55) | 200 mg Lasmiditan - MEE (N=53) | MEE - Control (N=54) | Open Label Extension (N=477)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngeal cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/403 (0) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 1/413 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication overuse headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/403 (0) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 2/413 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0/403 (0) | 0/418 (0) | 1/416 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/403 (0) | 1/418 (1) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1/403 (1) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0/403 (0) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 1/413 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 100 Milligram (mg) Lasmiditan (N=485) | 200 mg Lasmiditan (N=486) | Main - Control (N=500) | 100 mg Lasmiditan - MEE (N=55) | 200 mg Lasmiditan - MEE (N=53) | MEE - Control (N=54) | Open Label Extension (N=477)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 12 (19) | 7 (9) | 3 (3) | 0 (0) | 4 (5) | 0 (0) | 9 (17)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness transitory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 9 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (17)
Vertigo (Ear and labyrinth disorders) | 45 (68) | 47 (79) | 7 (7) | 0 (0) | 4 (7) | 0 (0) | 51 (211)
Vertigo positional (Ear and labyrinth disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid skin dryness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Metamorphopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 2 (3) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 1 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10)
Pupillary reflex impaired (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 5 (5) | 9 (12) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (20)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 2 (2) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (6) | 11 (14) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 6 (9) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 9 (58)
Dry mouth (Gastrointestinal disorders) | 6 (9) | 11 (15) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 3 (3) | 6 (6) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 56 (69) | 71 (105) | 29 (34) | 6 (7) | 4 (6) | 4 (7) | 60 (153)
Paraesthesia oral (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (14)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 13 (14) | 18 (22) | 11 (13) | 0 (0) | 3 (4) | 1 (1) | 21 (27)
Asthenia (General disorders) | 23 (32) | 31 (51) | 3 (4) | 8 (10) | 9 (13) | 2 (2) | 26 (60)
Chest discomfort (General disorders) | 2 (4) | 4 (7) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 3 (6)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 5 (6) | 5 (5) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 8 (19)
Discomfort (General disorders) | 5 (6) | 7 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (15)
Fatigue (General disorders) | 55 (80) | 71 (104) | 19 (21) | 3 (4) | 4 (6) | 2 (2) | 65 (241)
Feeling abnormal (General disorders) | 9 (9) | 19 (25) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Feeling cold (General disorders) | 6 (11) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling drunk (General disorders) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Feeling hot (General disorders) | 2 (4) | 6 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Feeling of body temperature change (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of relaxation (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (46)
Gait disturbance (General disorders) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 6 (9) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Non-cardiac chest pain (General disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 5 (7)
Sensation of blood flow (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sense of oppression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1/403 (1) | 1/418 (1) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 8 (8) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (14)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strength abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulse abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Food craving (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 8 (12) | 8 (11) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 12 (74)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 6 (17)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 (5) | 6 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (15)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 23 (36) | 29 (45) | 2 (3) | 6 (12) | 7 (10) | 1 (1) | 11 (39)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/403 (0) | 0/418 (0) | 1/416 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allodynia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 10 (15) | 13 (15) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 16 (43)
Bradykinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clumsiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (9)
Depressed level of consciousness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 7 (9) | 11 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Dizziness (Nervous system disorders) | 155 (230) | 187 (325) | 44 (59) | 24 (41) | 31 (61) | 6 (8) | 159 (770)
Dizziness postural (Nervous system disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysstasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fine motor skill dysfunction (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Formication (Nervous system disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 5 (20)
Headache (Nervous system disorders) | 9 (9) | 9 (10) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 18 (49)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 24 (33) | 16 (24) | 7 (9) | 3 (6) | 1 (2) | 1 (4) | 15 (30)
Hypotonia (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 5 (6) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (11)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mental impairment (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 72 (103) | 93 (170) | 21 (25) | 0 (0) | 3 (7) | 0 (0) | 72 (386)
Presyncope (Nervous system disorders) | 2 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (11)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 3 (6) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (40)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sedation (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensorimotor disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sensory disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Slow speech (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 32 (48) | 54 (82) | 12 (12) | 5 (7) | 10 (13) | 1 (2) | 49 (202)
Speech disorder (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 2 (2) | 1 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 8 (8) | 13 (21) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 16 (47)
Abnormal dreams (Psychiatric disorders) | 5 (5) | 6 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (32)
Aggression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 6 (8) | 10 (11) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 20 (47)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Daydreaming (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 3 (4) | 7 (8) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 6 (18)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (10)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Derealisation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorganised speech (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (17)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dyssomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 2 (2) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 2 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypnagogic hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (8) | 11 (20) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 15 (37)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 2 (4) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (15)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 3 (3) | 6 (9) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Sleep disorder (Psychiatric disorders) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 6 (6)
Somatic symptom disorder (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix inflammation (Reproductive system and breast disorders) | 0/403 (0) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 1/40 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/403 (1) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 2/413 (2)
Endometriosis (Reproductive system and breast disorders) | 0/403 (0) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 1/413 (1)
Erection increased (Reproductive system and breast disorders) | 0/82 (0) | 1/68 (1) | 0/84 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/403 (0) | 0/418 (0) | 1/416 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1/403 (1) | 0/418 (0) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 1/413 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0/403 (0) | 1/418 (1) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0/403 (0) | 0/418 (0) | 1/416 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/403 (0) | 1/418 (1) | 0/416 (0) | 0 (0) | 0 (0) | 0 (0) | 1/413 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 6 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Antibiotic prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth restoration (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 3 (6) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT03670810/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT03670810/SAP_001.pdf